CLINICAL TRIAL: NCT06205901
Title: A Prospective Comparison Study Between 18F-FDG PET/CT and Whole-Body Diffusion Weighted MRI in the Detection of Distant Malignancies in Patients With Various Cancers
Brief Title: Comparison Study Between PET/CT and Whole-Body Diffusion Weighted MRI in the Detection of Distant Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hala Mohamed Ahmed, Assistant lecturer, Radiology department, Sohag University
Other Study IDs: PET-CT and MRI in malignancy
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Distant Metastasis
Keywords: PET-CT, WB-MRI, Cancer patients, Distant metastasis
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET-CT, MRI — whole body MRI and PET-CT for cancer patients with distant metastasis

SUMMARY:
The purpose of the study is to compare the efficacy of 18F-FDG PET/CT and DWI WB-MRI in detection of distant metastasis of various cancers.

DETAILED DESCRIPTION:
Metastasis is the leading cause of morbidity and mortality in patients with cancer, accounting for ~90% of cancer-associated deaths.

Distant metastasis (DM) is a crucial point in the management of malignant tumors. DM is always associated with poor survival. Conclusive diagnosis of DM is crucial for improving the prognosis, reduction of the recurrence rate and hence, elevation of the 5-year survival rate.

Positron emission tomography/computed tomography (PET/CT) allows the analysis of active tumor tissue in the whole body. So, it obtains improved sensitivity and specificity when compared to conventional imaging modalities.

18F-FDG PET/CT is a diagnostic imaging modality with good quantitative properties. It has proven its interest in diagnosing, staging, and evaluating tumor response.

Whole-body MRI (WB-MRI) has been proposed as another effective whole-body approach for assessing both local invasiveness and distant metastases in patients with newly diagnosed cancers providing several advantages.

WB-MRI primarily provides structural information (revealing a detailed image of the pathology or lesion) on tumor spread; however, the absence of functional datasets has been resolved by incorporating Whole-body Diffusion Weighted Imaging (WB-DWI) into medical practice. WB-DWI shortens examination interpretation times by directing the radiologist's attention to abnormalities, which may then be investigated on anatomic sequences. It enables early detection of skeletal metastases as well as spread to other sites (liver and brain).

DW-MRI measures the Brownian motion of water molecules within intra- and extracellular spaces. This occurs in highly cellular lesions or in environments in which tissue architecture is disrupted and can be quantified by calculating the apparent diffusion coefficient (ADC).

ELIGIBILITY:
Inclusion Criteria:

* Only patients with malignancies proven by histology and patients with metastatic lesions proven by histopathology or cytology were included.

Exclusion Criteria:

* • As regard the PET/CT study, patients who have the general CT contraindications such as pregnancy, breast feeding, history of allergic reaction to the contrast medium, renal disease, etc.

  * As regard the MRI study, general contraindications including claustrophobia, MR-incompatible pacemakers and MR-incompatible heart valves.
  * Patients whose MRI sequences were incomplete, low-quality and/or had no histopathological evidence of metastatic lesions were eliminated from the study.
  * Low-quality or incomplete MRI included MRI exams with incomplete sequence(s), which is particularly common in elderly patients who are unable to tolerate the scan, or uncooperative patients who do not obey breathing instructions and motion artifacts that may impair images and lead to lower accuracy.
  * Declined consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patient, having present history of malignancy and referred from the general surgery or oncology clinics as having known metastatic lesions proven by histopathology or cytology. all Patients should be eligible to go through both modalities; PET-CT and MRI.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
comparison between the efficacy of 18F-FDG PET/CT and DWI WB-MRI in detection of distant metastasis of various cancers | 1 Year
  comparing the value of both PET-CT and whole body MRI mainly the DWI sequence in detection of bony and soft tissue metastasis in different types of malignancy. Which? will be better in early detection.
  PET-CT:
  differentiation of benign from malignant lesions can be determined using (Standardized uptake value) (SUV) as malignant lesions show higher SUV than benign lesions.
  Typically, a standardized uptake value (SUV) is a descriptive name of the quantity that incorporates the patient's size and the injected dose; > 2.0: considered malignancy, less than this value: considered to be benign.
  DWI WB-MRI:
  differentiation of benign from malignant lesions can be determined using ADC value as malignant lesions show low ADC value compared to the benign lesions.
  Apparent diffusion coefficient (ADC) is a descriptive name of the measure of the magnitude of diffusion (of water molecules) within tissue.

SECONDARY OUTCOMES:
DWI-MRI in detection of metastatic lesions in cancer patients | 1 Year
  detection of malignancy with applying ADC cut-off level for differentiating the malignant metastatic deposits.
  qualitative interpretation: differentiation of benign from malignant lesions can be determined through presence Vs absence diffusion restriction at diffusion weighted images (DWI), as only the malignant lesions that show diffusion restriction .
  quantitative interpretation: differentiation of benign from malignant lesions can be determined using ADC value as malignant lesions show low ADC value compared to the benign lesions.
  Apparent diffusion coefficient (ADC) is a descriptive name of the measure of the magnitude of diffusion (of water molecules) within tissue.
MRI in detection of metastatic lesions in cancer patients | 1 Year
  comparing each sequence of MRI in different organs including T2WI, T1WI and DWI sequences. ? Which is the best for detection and characterization of the Metastatic lesions in different bony and soft tissue in different parts of the body.
  T2WI & T1WI are descriptive names of sequences in the MRI study that can be evaluated qualitatively.
  DWI is a descriptive name of sequences in the MRI study that can be evaluated qualitatively and quantitively through using the ADC value which is a descriptive name of the measure of the magnitude of diffusion (of water molecules) within tissue.
Added value PET-CT in detection of metastatic lesions in cancer patients | 1 Year
  value of PET CT in detection of malignant metastatic deposits in bony and soft tissue lesions and the different pitfalls including the inflammatory conditions. Does the PET-CT can overcome it and how much sensitivity it has? qualitative interpretation : differentiation of benign from malignant lesions can be determined through the degree of 16F-FGD uptake as malignant lesions show avid uptake.
  quantitative interpretation: differentiation of benign from malignant lesions can be determined using (Standardized uptake value) (SUV) as malignant lesions show higher SUV than benign lesions.
  Typically, a standardized uptake value (SUV) is a descriptive name of the quantity that incorporates the patient's size and the injected dose, that is more than 2.0 is considered to be suggestive of malignancy, whereas lesions with SUVs less than this value are considered to be benign.
Accuracy of SUV value in PET-CT for detection of metastatic lesions in cancer patients | 1 Year
  detection of malignancy by applying Cut-Off level SUV value in detection and differentiation of metastatic deposits.

REFERENCES:
- [Background] Feng Y, Wang P, Chen Y, Dai W. 18 F-FDG PET/CT for evaluation of metastases in nonsmall cell lung cancer on the efficacy of immunotherapy. Nucl Med Commun. 2023 Oct 1;44(10):900-909. doi: 10.1097/MNM.0000000000001737. Epub 2023 Jul 31. PMID 37503694
- [Background] Rashid RJ, Tahir SH, Kakamad FH, Omar SS, Salih AM, Ahmed SF, Abdalla SH, Naqar S, Salih RQ, Kakamad SH, Mohammed KK, Mustafa SM, Hassan MN, Mohammed SH. Whole-body MRI for metastatic workup in patients diagnosed with cancer. Mol Clin Oncol. 2023 Mar 1;18(4):33. doi: 10.3892/mco.2023.2629. eCollection 2023 Apr. PMID 36925744
- [Background] Cristo Santos J, Henriques Abreu M, Seoane Santos M, Duarte H, Alpoim T, Prospero I, Sousa S, Henriques Abreu P. Bone Metastases Detection in Patients with Breast Cancer: Does Bone Scintigraphy Add Information to PET/CT? Oncologist. 2023 Aug 3;28(8):e600-e605. doi: 10.1093/oncolo/oyad087. PMID 37029988
- [Result] Chen J, Wu L, Zhang Z, Zheng S, Lin Y, Ding N, Sun J, Shi L, Xue M. A clinical model to predict distant metastasis in patients with superficial gastric cancer with negative lymph node metastasis and a survival analysis for patients with metastasis. Cancer Med. 2021 Feb;10(3):944-955. doi: 10.1002/cam4.3680. Epub 2020 Dec 22. PMID 33350173
- See also: Imaging in metastatic breast cancer, CT, PET/CT, MRI, WB-DWI, CCA: review and new perspectives — https://cancerimagingjournal.biomedcentral.com/articles/10.1186/s40644-023-00557-8#citeas
- See also: Detection of cancer before distant metastasis — https://bmccancer.biomedcentral.com/articles/10.1186/1471-2407-13-283